CLINICAL TRIAL: NCT02528604
Title: Cardioversion, Ablation or Pace and Ablate for Persistent Atrial Fibrillation in Over 65s - The CAPAPAF-65 Study
Brief Title: Electrical Cardioversion, Ablation or Pace and Ablate for Persistent Atrial Fibrillation
Acronym: CAPAPAF-65
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Principal Investigator, Rick Veasey, Consultant Cardiologist, Eastbourne General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPAPAF-65 V2.0
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Catheter Ablation; Permanent pacemaker; AV node ablation; Electrical Cardioversion; Implantable loop recorder
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Catheter Ablation (Active Comparator): Left atrial catheter ablation for persistent atrial fibrillation and implantable loop recorder.
  Interventions: Procedure: Catheter ablation; Device: Implantable loop recorder
- Pacemaker and AV node ablation (Active Comparator): Participants will have a permanent pacemaker implant followed by AV node ablation
  Interventions: Procedure: Pacemaker and AV node ablation
- DC cardioversion (Active Comparator): Participants will have electrical cardioversion with concomitant anti-arrhythmic therapy and implantable loop recorder.
  Interventions: Procedure: DC Cardioversion; Device: Implantable loop recorder

INTERVENTIONS:
Procedure: Catheter ablation — Left atrial ablation of persistent atrial fibrillation and implantable loop recorder insertion.
  Arms: Catheter Ablation
Procedure: Pacemaker and AV node ablation — Permanent pacemaker implant followed by AV node ablation
  Arms: Pacemaker and AV node ablation
Procedure: DC Cardioversion — Electrical cardioversion for Persistent Atrial Fibrillation and implantable loop recorder insertion.
  Arms: DC cardioversion
Device: Implantable loop recorder
  Arms: Catheter Ablation; DC cardioversion

SUMMARY:
Comparison of (i) catheter ablation, (ii) electrical cardioversion and (iii) pacemaker implantation with AV node ablation for patients over 65 years of age with persistent Atrial Fibrillation.

DETAILED DESCRIPTION:
the National Institute for Health and Care Excellence (NICE) suggest the following treatments options can be considered for patients with recurrent persistent atrial fibrillation:

1. Direct current cardioversion (DCCV) with concomitant anti-arrhythmic treatment.
2. Permanent pacemaker implantation (PPM) and atrio-ventricular (AV) node ablation.
3. Left atrial catheter ablation.

These treatment options have not been directly compared and each has their own advantages and disadvantages.

1. DC cardioversion is highly successful at restoring sinus rhythm and is a relatively cheap intervention. There is however a high recurrence rate of AF and cardioversion may need to be repeated multiple times.
2. Permanent pacemaker implantation and AV node ablation, 'ablate and pace' therapy provides rapid relief of symptoms and improved quality of life. Patients remain in atrial fibrillation but have a regular heart rhythm and controlled rate and avoid potential side-effects of medications. Following AV node ablation patients are dependent on the pacemaker and as such this treatment option is usually reserved for those over 65 years or age. Costs are modest and both the pacemaker insertion and AV node ablation procedures take less than 1 hour to perform.
3. Catheter ablation for atrial fibrillation aims to restore and sustain sinus rhythm. Procedural success rates are 50-60% after a single procedure and 80-85% after repeat procedures and it can take several months for all procedures in an ablation strategy to be performed. Procedural costs are high due to the equipment used and time taken for each ablation, usually 1.5-4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic persistent atrial fibrillation of less than 1-year duration.
* Patients must be over 65 years old.
* Patients give informed consent prior to participating in this study.

Exclusion Criteria:

* Paroxysmal atrial fibrillation.
* Long-standing persistent or permanent atrial fibrillation.
* Previous pacemaker implantation.
* Previous atrial ablation.
* Patient is unable to take warfarin or other oral anti-coagulant medication.
* Patient is suffering with unstable angina in last one week.
* Patient has had a myocardial infarction within last two months.
* Patient is expecting or has had major cardiac surgery within last two months.
* Patient is participating in a conflicting study.
* Patient is unable to perform exercise testing.
* Patient is mentally incapacitated and cannot consent or comply with follow-up.
* Patient has New York Heart Association (NYHA) class III/IV heart failure.
* Patient has left ventricular ejection fraction (LVEF) less than 35% not secondary to tachycardia.
* Pregnancy.
* Patient suffers with other cardiac rhythm disorders.
* Recent coronary artery intervention or other factors suggesting clinical instability (ECG, clinical or laboratory findings).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
AF recurrence | 12 months
  Time to recurrence of persistent AF

SECONDARY OUTCOMES:
Patient experience of procedure | Baseline
  Patient experience of each procedure will be assessed by validated questionnaires
Total costs of the treatment options | 12 months
AF recurrence >2minutes | 12 months
  Time to recurrence of AF episode > 2 minutes
Symptoms / QOL | 12 months
  To assess differences in symptoms and QOL
Exercise performance | 12 months
  To measure the three treatment effects on VO2 max over time by means of cardiopulmonary exercise testing.
AF burden | 12 months
  To measure the three treatment effects on AF burden
Sleep apnoea | 6 months
  To assess the impact of the three treatment options on sleep apnoea scores

CONTACTS AND LOCATIONS:
Overall Officials: Rick A Veasey, MRCP, MD, Principal Investigator — Consultant Cardiologist
Locations (2):
- United Kingdom (2):
  - Eastbourne District General Hospital, Eastbourne, East Sussex
  - Conquest Hospital, Saint Leonards-on-Sea, East Sussex